CLINICAL TRIAL: NCT03096418
Title: Neoadjuvant Weekly Paclitaxel and Biomarkers of Therapy Response
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16106; NCI-2017-00338 (Registry Identifier: NCI CTRP); 2016-1489 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 10/10/2025 (Other: UW Madison); 1R01CA284747-01A1 (NIH)
Record Dates: First submitted 2017-03-16; First posted 2017-03-30 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Weekly Paclitaxel (Experimental): Paclitaxel 80 mg/m2 will be initiated as standard infusion on days 1, 8, 15 of a 21-day cycle.
  Participants will continue with paclitaxel 80 mg/m2 for cycles 2-4 prior to surgery.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel is an FDA approved medication for treatment of curable breast cancer and is available by prescription at pharmacies throughout the United States.
  Other Names: Taxol

SUMMARY:
The hypothesis of this study is that paclitaxel levels increase chromosomal instability (CIN) in tumors and this is lethal to tumors that have pre-existing CIN. Treatment will be administered on an outpatient basis. Paclitaxel will be initiated as standard infusions on days 1, 8, and 15 of a 21-day cycle. Participants will continue with paclitaxel for cycles 2-4 prior to surgery.

DETAILED DESCRIPTION:
Primary Objectives

* To test if cancers with high chromosomal instability (CIN) respond to paclitaxel better than low CIN cancers.

Secondary Objectives

* To identify patient-specific differences in tumor levels and distribution of paclitaxel at 20 hours after first dose and patient-specific differences in peripheral non-tumor tissue (skin or plasma) paclitaxel levels 20 ± 4 hours after first dose.
* To determine if paclitaxel levels are higher at 20h after the 3rd dose than after the first dose, and if levels are higher at 20h after the 10th, 11th, or 12th dose than the 1st and 3rd dose.
* Compare pre-existing versus post-treatment antimitotic effects at 20h after the 1st dose, 20h after the 3rd dose, and 20h after the 10th, 11th, or 12th dose.
* Correlate drug levels and distribution with biomarkers including mitotic index, aneuploidy, chromosomal instability, and Ki67.
* Correlate pathologic response and clinical response with biomarkers including mitotic index, aneuploidy, CIN and Ki67.
* To test if CIN increases in patient tumors in response to paclitaxel and to evaluate the feasibility of these measurements by genomic analysis.

Initial Actual Primary and Study Completion Date registered as 8/16/2022 with 24 participants enrolled.

Per a Protocol Amendment dated 5/7/24, this study will re-open to enroll up to 50 participants. NCI funding and data sharing information added.

ELIGIBILITY:
Inclusion Criteria:

* Women with pathologically demonstrated breast cancer
* Patients must be candidates for neoadjuvant paclitaxel chemotherapy by their treating oncologist. No other investigational or commercial therapeutic agents may be given concurrently with the paclitaxel.
* Patients must not have metastatic disease on staging work-up per institutional guidelines.
* A formalin-fixed paraffin embedded tumor block (preferred) or unstained slides must be available from a prior biopsy of the primary tumor (preferred) or lymph node. A minimum of 8 slides must be available.
* The primary tumor or lymph node must be readily biopsied by surgery or radiology teams.
* The primary tumor must be measurable by an imaging modality prior to treatment. This imaging modality is to be repeated after completion of 4 cycles of paclitaxel and prior to surgery. Such imaging modalities may include ultrasound, CT, mammography, or MRI. MRI will be the preferred imaging modality if available because it has the highest accuracy and positive predictive value for predicting pathologic complete response.All imaging will be performed per standard of care at the discretion of the treating physicians.
* Subjects may not have had prior systemic chemotherapy regimens administered for treatment of their current breast cancer. However, studies (window studies, for example) that are deemed non-therapeutic, including those that utilize agents that are not FDA approved for the treatment of the patient's current breast cancer, are permitted.
* Patients must have adequate organ and marrow function as determined by the treating oncologist.
* Patient must be willing to undergo additional biopsy of breast tumor or lymph node.
* Patient must have the ability and willingness to sign a written informed consent document.
* Women of childbearing potential (per institutional policy) must agree to use effective contraception as discussed with treating oncologist for the duration of the study.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel including to other drugs formulated in Cremophor(R) EL (polyoxyethylated castor oil).
* Patients with known HIV due to concern that chemotherapy may cause further immunosuppression and potential infectious complications.
* Patients on non-aspirin anti-coagulation (Coumadin, heparins, or clopidogrel) or with documented bleeding disorders will be excluded due to risk of bleeding with biopsy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active severe infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, other malignancies requiring therapy or psychiatric illness/social situations that would limit compliance with study requirements as determined by treatment physician.
* Pregnant women are excluded from this study because paclitaxel is a pregnancy category D drug and may cause deleterious effects to the fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with paclitaxel, breastfeeding should be discontinued if the mother is enrolled in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Sharifi, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Iowa Health Care/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Scribano CM, Wan J, Esbona K, Tucker JB, Lasek A, Zhou AS, Zasadil LM, Molini R, Fitzgerald J, Lager AM, Laffin JJ, Correia-Staudt K, Wisinski KB, Tevaarwerk AJ, O'Regan R, McGregor SM, Fowler AM, Chappell RJ, Bugni TS, Burkard ME, Weaver BA. Chromosomal instability sensitizes patient breast tumors to multipolar divisions induced by paclitaxel. Sci Transl Med. 2021 Sep 8;13(610):eabd4811. doi: 10.1126/scitranslmed.abd4811. Epub 2021 Sep 8. PMID 34516829
- See also: UW Carbone Cancer Center Home Page — http://www.uwhealth.org/uw-carbone-cancer-center/cancer/10252

RESULTS

PARTICIPANT FLOW:
Groups:
- Weekly Paclitaxel: Paclitaxel 80 mg/m2 will be initiated as standard infusion on days 1, 8, 15 of a 21-day cycle.
  Participants will continue with paclitaxel 80 mg/m2 for cycles 2-4 prior to surgery.
  Paclitaxel: Paclitaxel is an FDA approved medication for treatment of curable breast cancer and is available by prescription at pharmacies throughout the United States.
Period: Overall Study
Arm/Group | Weekly Paclitaxel
Started | 24
Paclitaxel Concentration Determine | 15
Analyzed After First Dose | 16
Analyzed After Third Dose | 5
Analyzed After Twelfth Dose | 1
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Weekly Paclitaxel
Number analyzed (Participants) | 24
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1
  30-39 years | 4
  40-49 years | 7
  50-59 years | 7
  60-69 years | 2
  70-79 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Response to Paclitaxel
Description: To test if high cancers with high chromosomal instability (CIN) respond to paclitaxel better than low CIN cancers. Response determined by the percent decrease in linear measurement of tumor size on the greatest dimension per RECIST-like criteria
Time Frame: Up to 3 months
Population: Only 12 participants were evaluable because of insufficient specimen.
Measure: Mean (Full Range); unit: percent decrease in tumor size
Arm/Group | Weekly Paclitaxel
Number analyzed (Participants) | 12
percent decrease in tumor size | -29.63 [-70.21 to 30]

2. Secondary Outcome: Tumor Level Difference of Paclitaxel
Description: Identify patient-specific differences in tumor levels of paclitaxel at 20 hours after first dose.
  This is measured by high-performance liquid chromatography of tumor and plasma samples and comparing variability between patients with descriptive statistics.
Time Frame: Up to 1 day
Population: Participant 10 withdrew consent.
Measure: Number; unit: micromolar
Arm/Group | Weekly Paclitaxel
Number analyzed (Participants) | 14
micromolar
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 1.07
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 0.34
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 0.80
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 0.57
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 3.43
  Participant 7: number analyzed (Participants) | 1
  Participant 7 | 1.55
  Participant 8: number analyzed (Participants) | 1
  Participant 8 | 0.53
  Participant 9: number analyzed (Participants) | 1
  Participant 9 | 0.63
  Participant 11: number analyzed (Participants) | 1
  Participant 11 | 0.57
  Participant 13: number analyzed (Participants) | 1
  Participant 13 | 1.67
  Participant 14: number analyzed (Participants) | 1
  Participant 14 | 0.52
  Participant 15: number analyzed (Participants) | 1
  Participant 15 | 1.20
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | NA — Insufficient tumor tissue collected by biopsy
  Participant 12: number analyzed (Participants) | 1
  Participant 12 | NA — Insufficient tumor tissue collected by biopsy

3. Secondary Outcome: Non-Tumor Level Difference of Paclitaxel
Description: Identify patient-specific differences in non-tumor (plasma) levels of paclitaxel at 20 hours after first dose.
  This is measured by high-performance liquid chromatography of tumor and plasma samples and comparing variability between patients with descriptive statistics.
Time Frame: Up to 1 day
Population: Participant 10 withdrew consent
Measure: Number; unit: micromolar
Arm/Group | Weekly Paclitaxel
Number analyzed (Participants) | 14
micromolar
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 0.023
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 0.040
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 0.030
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 0.027
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 0.031
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 0.020
  Participant 7: number analyzed (Participants) | 1
  Participant 7 | 0.013
  Participant 8: number analyzed (Participants) | 1
  Participant 8 | 0.011
  Participant 9: number analyzed (Participants) | 1
  Participant 9 | 0.020
  Participant 11: number analyzed (Participants) | 1
  Participant 11 | 0.038
  Participant 12: number analyzed (Participants) | 1
  Participant 12 | 0.040
  Participant 13: number analyzed (Participants) | 1
  Participant 13 | 0.094
  Participant 14: number analyzed (Participants) | 1
  Participant 14 | 0.048
  Participant 15: number analyzed (Participants) | 1
  Participant 15 | 0.035

4. Secondary Outcome: Paclitaxel Levels
Description: Paclitaxel levels at the first dose, 20 hours after the 3rd dose, and 20 hours after the 12th dose. This is measured by high-performance liquid chromatography of tumor and plasma samples and comparing difference at two time points within the same patient with paired statistics.
Time Frame: Up to 79 days
Measure: Mean (Full Range); unit: micromolars
Arm/Group | Weekly Paclitaxel
Number analyzed (Participants) | 7
micromolars
  First dose plasma paclitaxel | 0.041 [0.014 to 0.094]
  Third dose plasma paclitaxel | 0.029 [0.013 to 0.062]
  First dose intratumoral paclitaxel | 0.785 [0.34 to 1.67]
  Third dose intratumoral paclitaxel | 1.21 [0.12 to 2.40]

5. Secondary Outcome: Antimitotic Effects
Description: Compare pre-existing versus post-treatment antimitotic effects at 20 hours after the 1st dose, 20 hours after the 3rd dose, and 20 hours after the 12th dose.
  This is measured by tissue analysis of tumor samples with phospho-histone H3 and stains for spindle morphology to quantify mitotic index and mitotic characteristics at two time points using paired statistical analysis.
Time Frame: Up to 79 days
Population: An increasing smaller subset of participants were biopsied after the first dose.
Measure: Number; unit: number of mitotic cells
Groups:
- Weekly Paclitaxel - Baseline; Weekly Paclitaxel - 20 Hours After First Dose; Weekly Paclitaxel - 20 Hours After Third Dose; Weekly Paclitaxel - 20 Hours After Twelfth Dose: Paclitaxel 80 mg/m2 will be initiated as standard infusion on days 1, 8, 15 of a 21-day cycle.
  Participants will continue with paclitaxel 80 mg/m2 for cycles 2-4 prior to surgery.
  Paclitaxel: Paclitaxel is an FDA approved medication for treatment of curable breast cancer and is available by prescription at pharmacies throughout the United States.
Arm/Group | Weekly Paclitaxel - Baseline | Weekly Paclitaxel - 20 Hours After First Dose | Weekly Paclitaxel - 20 Hours After Third Dose | Weekly Paclitaxel - 20 Hours After Twelfth Dose
Number analyzed (Participants) | 16 | 16 | 5 | 1
number of mitotic cells
  Participant 1: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 1 | 113 | 109 |  |
  Participant 2: number analyzed (Participants) | 1 | 1 | 1 | 0
  Participant 2 | 41 | 100 | 32 |
  Participant 3: number analyzed (Participants) | 1 | 1 | 1 | 0
  Participant 3 | 100 | 104 | 105 |
  Participant 4: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 4 | 101 | 103 |  |
  Participant 6: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 6 | 106 | 108 |  |
  Participant 7: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 7 | 79 | 103 |  |
  Participant 8: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 8 | 75 | 27 |  |
  Participant 9: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 9 | 35 | 63 |  |
  Participant 11: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 11 | 6 | 11 |  |
  Participant 12: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 12 | 24 | 30 |  |
  Participant 13: number analyzed (Participants) | 1 | 1 | 1 | 0
  Participant 13 | 106 | 110 | 101 |
  Participant 14: number analyzed (Participants) | 1 | 1 | 1 | 0
  Participant 14 | 86 | 102 | 20 |
  Participant 15: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 15 | 116 | 101 |  |
  Participant 16: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 16 | 106 | 104 |  |
  Participant 18: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 18 | 42 | 214 | 23 | 8
  Participant 19: number analyzed (Participants) | 1 | 1 | 0 | 0
  Participant 19 | 30 | 70 |  |

6. Secondary Outcome: Mitotic Index
Description: The mitotic index is a measure of cells arresting in mitosis, previously thought to be the major mechanism of taxol action. It is defined as the percentage of cells undergoing mitosis in a given population of cells. An elevated mitotic index indicates more cells are at this phase of the cell cycle at the time of sampling.
Time Frame: Baseline and 20 hours post-first dose
Population: Clinical Response reported here.
Measure: Number; unit: mitotic index
Groups:
- Weekly Paclitaxel - Pre-treatment; Weekly Paclitaxel - 20 Hours Post-first Dose: Paclitaxel 80 mg/m2 will be initiated as standard infusion on days 1, 8, 15 of a 21-day cycle.
  Participants will continue with paclitaxel 80 mg/m2 for cycles 2-4 prior to surgery.
  Paclitaxel: Paclitaxel is an FDA approved medication for treatment of curable breast cancer and is available by prescription at pharmacies throughout the United States.
Arm/Group | Weekly Paclitaxel - Pre-treatment | Weekly Paclitaxel - 20 Hours Post-first Dose
Number analyzed (Participants) | 13 | 13
mitotic index
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 1.4 | 2.6
  Participant 2: number analyzed (Participants) | 1 | 1
  Participant 2 | 1 | 3.379722
  Participant 3: number analyzed (Participants) | 1 | 1
  Participant 3 | 1.35 | 4.4
  Participant 4: number analyzed (Participants) | 1 | 1
  Participant 4 | 1.8 | 3.192745
  Participant 6: number analyzed (Participants) | 1 | 1
  Participant 6 | 1.052765 | 2.305837
  Participant 7: number analyzed (Participants) | 1 | 1
  Participant 7 | 1.2 | 3.201638
  Participant 8: number analyzed (Participants) | 1 | 1
  Participant 8 | 0.6 | 1.29731
  Participant 9: number analyzed (Participants) | 1 | 1
  Participant 9 | 1.466667 | 1.872558
  Participant 11: number analyzed (Participants) | 1 | 1
  Participant 11 | 0.198311 | 0.32
  Participant 12: number analyzed (Participants) | 1 | 1
  Participant 12 | 0.32 | 1.44
  Participant 13: number analyzed (Participants) | 1 | 1
  Participant 13 | 2 | 4.2
  Participant 14: number analyzed (Participants) | 1 | 1
  Participant 14 | 1.48 | 2.87
  Participant 15: number analyzed (Participants) | 1 | 1
  Participant 15 | 1.33 | 5.56

7. Secondary Outcome: Correlate Drug Levels With Aneuploidy of Tumor
Description: Correlate pathologic response and clinical response with biomarkers including aneuploidy
Time Frame: Up to 3 months
Population: This biomarker was not measured
Arm/Group | Weekly Paclitaxel
Number analyzed (Participants) | 0

8. Secondary Outcome: Correlate Drug Levels With Chromosomal Instability of Tumor
Description: Correlate pathologic response and clinical response with biomarkers including CIN
Time Frame: Up to 3 months
Population: This was not measured
Arm/Group | Weekly Paclitaxel
Number analyzed (Participants) | 0

9. Secondary Outcome: Ki67 of Tumor
Description: The Ki-67 protein is a cellular marker for proliferation. Ki-67 is an excellent marker to determine the growth fraction of a given cell population. The fraction of Ki-67-positive tumor cells (the Ki-67 labeling index) is often correlated with the clinical course of cancer.
Time Frame: Up to 3 months
Population: Clinical Response reported here.
Measure: Number; unit: Percentage of Ki67 + cells
Arm/Group | Weekly Paclitaxel
Number analyzed (Participants) | 12
Percentage of Ki67 + cells
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 90
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 80
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 90
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 45
  Participant 7: number analyzed (Participants) | 1
  Participant 7 | 90
  Participant 8: number analyzed (Participants) | 1
  Participant 8 | 60
  Participant 9: number analyzed (Participants) | 1
  Participant 9 | 15
  Participant 11: number analyzed (Participants) | 1
  Participant 11 | 20
  Participant 12: number analyzed (Participants) | 1
  Participant 12 | 25
  Participant 13: number analyzed (Participants) | 1
  Participant 13 | 90
  Participant 14: number analyzed (Participants) | 1
  Participant 14 | 60
  Participant 15: number analyzed (Participants) | 1
  Participant 15 | 60

10. Secondary Outcome: Change in CIN Levels
Description: There are many proposed ways to measure CIN. Here, we used # of multipolar spindles as a surrogate of CIN measures.
Time Frame: Baseline and 20 hours post-first dose
Population: Insufficient tissue was collected to complete analysis on remaining participants
Measure: Number; unit: % of cells with multipolar spindles
Groups:
- Weekly Paclitaxel Pre-treatment; Weekly Paclitaxel - 20 Hours After First Dose: Paclitaxel 80 mg/m2 will be initiated as standard infusion on days 1, 8, 15 of a 21-day cycle.
  Participants will continue with paclitaxel 80 mg/m2 for cycles 2-4 prior to surgery.
  Paclitaxel: Paclitaxel is an FDA approved medication for treatment of curable breast cancer and is available by prescription at pharmacies throughout the United States.
Arm/Group | Weekly Paclitaxel Pre-treatment | Weekly Paclitaxel - 20 Hours After First Dose
Number analyzed (Participants) | 13 | 13
% of cells with multipolar spindles
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 7.08 | 51.38
  Participant 2: number analyzed (Participants) | 1 | 1
  Participant 2 | 2.44 | 49
  Participant 3: number analyzed (Participants) | 1 | 1
  Participant 3 | 2.44 | 26.92
  Participant 4: number analyzed (Participants) | 1 | 1
  Participant 4 | 3.96039604 | 29.12621359
  Participant 6: number analyzed (Participants) | 1 | 1
  Participant 6 | 16.98113208 | 60.18518519
  Participant 7: number analyzed (Participants) | 1 | 1
  Participant 7 | 3.797468354 | 64.0776699
  Participant 8: number analyzed (Participants) | 1 | 1
  Participant 8 | 5.33333333 | 62.96296296
  Participant 9: number analyzed (Participants) | 1 | 1
  Participant 9 | 8.571428571 | 61.9047619
  Participant 11: number analyzed (Participants) | 1 | 1
  Participant 11 | 0 | 27.27
  Participant 12: number analyzed (Participants) | 1 | 1
  Participant 12 | 4.2 | 56.6
  Participant 13: number analyzed (Participants) | 1 | 1
  Participant 13 | 5.6 | 64.5
  Participant 14: number analyzed (Participants) | 1 | 1
  Participant 14 | 13.95 | 58.82
  Participant 15: number analyzed (Participants) | 1 | 1
  Participant 15 | 3.45 | 60.4

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Weekly Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03096418/Prot_SAP_000.pdf